CLINICAL TRIAL: NCT04714697
Title: Cabozantinib as Subsequent Therapy to an Immune Checkpoint Based Therapy in Renal Cell Carcinoma, Phase 2, Interventional Study
Brief Title: Cabozantinib as Subsequent Therapy to an Immune Checkpoint Based Therapy in Renal Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Principal Investigator, Jae-Lyun Lee, professor, Asan Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AT ASIA
Record Dates: First submitted 2021-01-07; First posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1(post nivolumab and ipilimumab combination) (Experimental): the subject who failed one prior line by nivolumab and ipilimumab
  Interventions: Drug: Cabometyx
- Cohort 2 (post pembrolizumab plus axitinib, pembrolizumab plus lenvatinib, or avelumab and axitinib) (Experimental): the subject who failed one prior line by PD-1/PD-L1 inhibitors in combination with VEGF TKI
  Interventions: Drug: Cabometyx
- Cohort 3 (post sequential immunotherapy after VEGFR TKI) (No Intervention): the subject who failed the second line by immunotherapy (PD-1 antibody or PD-L1 antibody) following the first line VEGFR TKI

INTERVENTIONS:
Drug: Cabometyx — Cabometyx 60mg once daily, oral , up to Progression disease
  Arms: Cohort 1(post nivolumab and ipilimumab combination); Cohort 2 (post pembrolizumab plus axitinib, pembrolizumab plus lenvatinib, or avelumab and axitinib)

SUMMARY:
This study is a phase 2, multicenter, interventional for cohort 1 & 2, non-interventional for cohort 3, open-label trial of cabozantinib, with ORR as the primary efficacy endpoint. In total, 201 eligible subjects will enroll from 5 sites in Korea. The intervention for this cohort 1&2 is only IMP, Cabometyx provided by Ipsen (off-label). Also, cohort 3 is just RWD without IMP (on-label)

DETAILED DESCRIPTION:
Cohort 1 (post nivolumab and ipilimumab combination): the subject who failed one prior line by nivolumab and ipilimumab Cohort 2 (post pembrolizumab plus axitinib, pembrolizumab plus lenvatinib, or avelumab and axitinib): the subject who failed one prior line by PD-1/PD-L1 inhibitors in combination with VEGF TKI Cohort 3 (post sequential immunotherapy after VEGFR TKI): the subject who failed the second line by immunotherapy (PD-1 antibody or PD-L1 antibody) following the first line VEGFR TKI Subjects will receive study treatment as long as they continue to experience a clinical benefit in the investigator's opinion or until there is unacceptable toxicity or the need for subsequent systemic anticancer therapy. Treatment may continue after radiographic progression per RECIST 1.1 as long as the investigator believes that the subject is still receiving clinical benefit from study treatment and that the potential benefit of continuing study treatment outweighs potential risks.

ELIGIBILITY:
Inclusion Criteria:

1. Documented histological or cytological diagnosis of advanced renal cell cancer with or without clear-cell component with an exception of collecting duct carcinoma
2. Measurable disease per RECIST 1.1, as determined by the investigator.
3. Recovery to baseline or/and under Grade 1 CTCAE v.5.0 from toxicities related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy.
4. Age eighteen years or older on the day of consent.
5. Karnofsky Performance Status (KPS) score of or/and over 70%.
6. Adequate organ and marrow function, based upon meeting all of the following laboratory criteria within ten days before randomization:
7. Capable of understanding and complying with the protocol requirements and must have signed the informed consent document.
8. Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception (e.g., barrier methods, including male condom, female condom).
9. Female subjects of childbearing potential must not be pregnant at the screening. Females of childbearing potential are defined as premenopausal females capable of becoming pregnant (i.e., females who have had any evidence of menses in the past 12 months, except for those who had a prior hysterectomy). However, women who have been amenorrheic for 12 or more months are still considered childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, low body weight,ovarian suppression, or other reasons.
10. Cohort-Specific Criteria Cohort 1

    1. Must have received nivolumab and ipilimumab combination as the first-line systemic treatment
    2. Subjects who experienced disease progression on nivolumab and ipilimumab combination or unacceptable toxicities.

Cohort 2

1. Must have received pembrolizumab plus axitinib, pembrolizumab plus Lenvatinib, or avelumab plus axitinib combination as the first-line systemic treatment
2. Subjects who experienced disease progression on PD-1/PD-L1 inhibitors with VEGFR TKI combination or unacceptable toxicities.

Cohort 3

1. Must have received VEGFR TKI (e.g., sunitinib, axitinib, pazopanib, or sorafenib) as the first-line systemic treatment and sequential PD-1 antibody or PD-L1 antibody, e.g., Pembrolizumab, nivolumab, atezolizumab, avelumab, durvalumab, PDR001.
2. Subjects who experienced disease progression on second-line PD-1 or PD-L1 antibody or unacceptable toxicities.

Exclusion Criteria:

1. Prior treatment with cabozantinib.
2. Treated with any other investigational medicinal product (IMP) within the last 30 days before screening
3. For cohort 1 & 2, concurrent involvement participation in any investigational study.
4. For cohort 3, participation in cabozantinib rPMS during the study
5. Radiation therapy for bone metastasis within one week, any other external radiation therapy within two weeks before randomization. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible.
6. Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least one month before randomization. Eligible subjects must be neurologically asymptomatic at the time of enrollment.
7. Concomitant anticoagulation at therapeutic doses with oral anticoagulants (e.g., warfarin, direct thrombin, and Factor Xa inhibitors) or platelet inhibitors (e.g., clopidogrel).

   Note: Low-dose aspirin for cardioprotection (per locally applicable guidelines), low-dose warfarin (under 1 mg/day), and low dose, low molecular weight heparins (LMWH) are permitted. Anticoagulation with therapeutic doses of LMWH is allowed in subjects without radiographic evidence of brain metastasis, who are on a stable dose of LMWH for at least 12 weeks before randomization, and who have had no complications from a thromboembolic event or the anticoagulation regimen.
8. The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

   1. Cardiovascular disorders:

      * Symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmias.
      * Uncontrolled hypertension defined as sustained BP above 150 mm Hg systolic or 100 mm Hg diastolic despite optimal antihypertensive treatment.
      * Stroke (including TIA), myocardial infarction, or other ischemic event, or thromboembolic event (eg, deep venous thrombosis, pulmonary embolism) within 6 months before randomization.
   2. Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:

      - Tumors invading the GI-tract, active peptic ulcer disease, inflammatory bowel disease, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis or acute obstruction of the pancreatic or biliary duct, or gastric outlet obstruction.

      Abdominal fistula, gastrointestinal perforation, bowel obstruction, or intra-abdominal abscess within 6 months before randomization.

      Note: Complete healing of an intra-abdominal abscess must be confirmed before randomization.
   3. Clinically significant hematuria, hematemesis, or hemoptysis of above 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (eg, pulmonary hemorrhage) within 3 months before enrollment.
   4. Cavitray lung lesions or documented endobronchial lesions
   5. Lesions invading major pulmonary blood vessels.
   6. Other clinically significant disorders such as:

      * Active infection requiring systemic treatment, infection with human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)- related illness.
      * Serious non-healing wound/ulcer/bone fracture.
      * Malabsorption syndrome.
      * Moderate to severe hepatic impairment (Child-Pugh B or C).
      * History of solid organ transplantation.
9. Major surgery (eg, GI surgery, removal or biopsy of brain metastasis) within 1 month before IP administration. Complete wound healing from major surgery or minor surgery (eg, simple excision, tooth extraction) must have occurred 1 month before IP administration. Subjects with clinically relevant ongoing complications from prior surgery are not eligible.
10. Corrected QT interval calculated by the Fridericia formula (QTcF) above 500 msec within 1 month before randomization (see Section 5.5.4 for Fridericia formula).

    Three ECGs must be performed. If the average of these three consecutive results for QTcF is or/and under 500 msec, the subject meets eligibility in this regard.
11. Pregnant or lactating females.
12. Inability to swallow tablets or capsules.
13. Previously identified allergy or hypersensitivity to components of the study treatment formulations.
14. Diagnosis of another malignancy within 1 year before randomization, except for superficial skin cancers, or localized, low grade tumors deemed cured and not treated with systemic therapy.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | up to 2years
  Objective response rate , per RECIST 1.1, per investigator assessment

SECONDARY OUTCOMES:
Time to response, | up to 2years
  Time to response, per RECIST 1.1, per investigator assessment
Duration of response | up to 2years
  Duration of response, per RECIST 1.1, per investigator assessment
Progression-free survival | up to 2years
  Progression-free survival , per RECIST 1.1, per investigator assessment
Overall survival | up to 5years
  Overall survival
Incidence of Treatment Adverse Events incidence of treatment Adverse Events (safety) | From date of Cycle 1Day 1 (first dosing) until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24months
  Adverse Event, Serious adverse event by CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shah AY, Kotecha RR, Lemke EA, Chandramohan A, Chaim JL, Msaouel P, Xiao L, Gao J, Campbell MT, Zurita AJ, Wang J, Corn PG, Jonasch E, Motzer RJ, Sharma P, Voss MH, Tannir NM. Outcomes of patients with metastatic clear-cell renal cell carcinoma treated with second-line VEGFR-TKI after first-line immune checkpoint inhibitors. Eur J Cancer. 2019 Jun;114:67-75. doi: 10.1016/j.ejca.2019.04.003. Epub 2019 May 7. PMID 31075726